CLINICAL TRIAL: NCT02654860
Title: Two-part Study of Intrathecal Paracetamol Administered Immediately Before Spinal Anaesthesia in Patients Scheduled for Hip Replacement Surgery
Brief Title: Dose-finding Study of Intrathecal Paracetamol Administered Immediately Before Spinal Anaesthesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Collaborators: Cross S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PAR.3/02-2015
Record Dates: First submitted 2015-12-23; First posted 2016-01-13 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-07

CONDITIONS: Phase 1: Pain Management; Phase 2: Pain Management
MeSH Terms: interventions — 3-(cystein-S-yl)paracetamol

STUDY DESIGN:
Intervention Model Description: 4 arms for Phase II only
Who Masked: Participant, Investigator
Masking Description: Phase II only
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 60 mg Paracetamol 3% (2 mL) (Experimental): 60 mg Paracetamol 3%. Solution for injection, single administration by Intrathecal route.
  Interventions: Drug: Paracetamol 3%; Drug: Hyperbaric Bupivacaine HCl 0.5%
- 90 mg Paracetamol 3% (3 mL) (Experimental): 90 mg Paracetamol 3%. Solution for injection, single administration by Intrathecal route.
  Interventions: Drug: Paracetamol 3%; Drug: Hyperbaric Bupivacaine HCl 0.5%
- 120 mg Paracetamol 3% (4mL) (Experimental): 120 mg Paracetamol 3%. Solution for injection, single administration by Intrathecal route.
  Interventions: Drug: Paracetamol 3%; Drug: Hyperbaric Bupivacaine HCl 0.5%
- Phase II Only: Saline solution 0.9% (Placebo Comparator): Placebo, 0.9%. Solution for injection , single administration by route Intrathecal (2 mL, 3 mL and 4 mL) Study part 2 will be placebo-controlled. Each patient will be allocated to a treatment arm (one of the three paracetamol doses or placebo) according to a computer-generated randomisation list.
  Interventions: Drug: Placebo injection containing Saline solution 0.9%; Drug: Hyperbaric Bupivacaine HCl 0.5%

INTERVENTIONS:
Drug: Paracetamol 3% — Investigate the efficacy and safety of a single intrathecal injection of paracetamol,for post-operative analgesia of hip replacement surgery
  Arms: 120 mg Paracetamol 3% (4mL); 60 mg Paracetamol 3% (2 mL); 90 mg Paracetamol 3% (3 mL)
Drug: Placebo injection containing Saline solution 0.9% — Injection containing sterile solution of Saline Solution 0.9 %. Study part 2 will be placebo-controlled. Each patient will be allocated to a treatment arm (one of the three paracetamol doses or placebo) according to a computer-generated randomisation list.
  Arms: Phase II Only: Saline solution 0.9%
Drug: Hyperbaric Bupivacaine HCl 0.5% — NIMP, spinal anaesthetic before the surgical procedure

SUMMARY:
Two-part study of intrathecal paracetamol administered immediately before spinal anaesthesia in patients scheduled for hip replacement surgery

DETAILED DESCRIPTION:
This is a prospective, single centre, two-part, three doses study. Part 1 is a Phase I, three cohorts, dose-ascending, open-label, safety study. Part 2 is a Phase II, randomised, parallel-group, double-blind, placebo-controlled, exploratory efficacy and safety study The objective of the study is to investigate the efficacy and safety of a single intrathecal injection of paracetamol, administered at 3 doses to 3 active treatment groups, as compared to placebo solution, for post-operative analgesia of hip replacement surgery performed under spinal anaesthesia. Patients scheduled for hip replacement surgery will be randomised into 4 treatment groups (15 patients per group) to receive either one of the 3 single doses of paracetamol 3% (D1: 60 mg, D2: 90 mg, D3: 120 mg) or placebo solution (P: saline solution) by intrathecal (IT) injection. Immediately after paracetamol or placebo IT administration, all patients will receive a single IT dose of Hyperbaric Bupivacaine HCl 0.5% (12.5 mg for ≤ 160 cm-tall patients and 15 mg for > 160 cm-tall patients). The time interval between paracetamol IT and bupivacaine IT administrations should not exceed 2 min.

The study will include a screening phase (Visit 1, Days -21/1), a treatment phase (paracetamol IT administration, anaesthesia and surgical procedure: Visit 2, Day 1) and a follow-up phase including an observation period (Visit 3, from Day 1 after surgery until discharge, a final visit (at discharge) and a follow-up (day 6±1). Pain at rest will be assessed at screening and on visit 2 at baseline (0 h), 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45 and 48 h after anaesthetic IT injection and at discharge, using a 0-100 mm VAS.

ELIGIBILITY:
Inclusion Criteria Phase 1 and Phase 2:

* Informed consent: signed written informed consent before inclusion in the study
* Sex, age and surgery: male/female 18-80 years (inclusive) old patients, scheduled for hip replacement surgery, with anticipated need for post-operative narcotic analgesia, adequate i.v. access and anticipated hospital stay > 48 hours.
* Body Mass Index (BMI): 18 - 34 kg/m2 inclusive
* ASA physical status: I-III
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
* Inclusion criteria - Phase 1 only : Age: 18-70 (inclusive) old patients
* Inclusion criteria - Phase 2 only : Age: 18-80 (inclusive) old patients Hospital stay: Patients with anticipated hospital stay > 48 hours

Exclusion Criteria Phase 1 and Phase 2:

* Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study. Contraindications to spinal anaesthesia. History of neuromuscular diseases to the lower extremities
* ASA physical status: IV-V
* Further anaesthesia: patients expected to require further anaesthesia
* Pain assessment: anticipated to be unable to make a reliable self-report of pain intensity
* Allergy: ascertained or presumptive hypersensitivity to the active principles (paracetamol and/or amide type anaesthetics) and/or formulations' ingredients or related drugs, opioids, non-steroidal anti-inflammatory drugs; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers could affect the outcome of the study
* Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; ascertained psychiatric and neurological diseases, sepsis, blood coagulation disorders, severe cardiopulmonary disease, thyroid disease, diabetes, other neuropathies, history or evidence of asthma or heart failure. History of severe head trauma that required hospitalisation, intracranial surgery or stroke within the previous 30 days, or any history of intracerebral arteriovenous malformation, cerebral aneurism or CNS mass lesion.
* Liver function: Impaired liver function (transaminases > twice upper limit)
* Renal function: Renal dysfunction (creatinine > 2.0 mg/dL)
* Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study, calculated from the first day of the month following the last visit of the previous study
* Drug, alcohol: history of drug or alcohol abuse. Pre-existing dependence on narcotics or known tolerance to opioids
* Pregnancy and lactation: positive pregnancy test at screening (if applicable), pregnant or lactating women [The pregnancy test will be performed to all fertile women and to all women up to 55 years old, if not in proven menopause (available laboratory test confirming menopause or surgically sterilised)]
* Chronic pain syndromes: patients with chronic pain syndromes (taking opioids, anticonvulsant agents or chronic analgesic therapy).
* Medications: medication known to interfere with the extent of spinal blocks for 2 weeks before the start of the study. Paracetamol formulations, other than the investigational product, for 1 week before the start of the study and during the study. Hormonal contraceptives for females are allowed.
* Phase 2 only - Exclusion criteria Pain assessment: anticipated to be unable to make a reliable self-report of pain intensity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-11; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Camponovo, MD, Principal Investigator — Department of Anaesthesiology,Clinica Ars Medica,Via Cantonale, CH-6929 Gravesano, Switzerland
Locations (1):
- Claudio Camponovo, Gravesano, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II Only: Saline Solution 0.9%: Placebo, 0.9%. Solution for injection , single administration by route Intrathecal (2 mL, 3 mL and 4 mL) Study part 2 will be placebo-controlled. Each patient will be allocated to a treatment arm (one of the three paracetamol doses or placebo) according to a computer-generated randomisation list.
  Placebo injection containing Saline solution 0.9%: Injection containing sterile solution of Saline Solution 0.9 %.
  Study part 2 will be placebo-controlled. Each patient will be allocated to a treatment arm (one of the three paracetamol doses or placebo) according to a computer-generated randomisation list.
  Hyperbaric Bupivacaine HCl 0.5%: NIMP, spinal anaesthetic before the surgical procedure
Period: First Part
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Started | 3 | 3 | 3 | 0
Completed | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Second Part
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9% | Total
Number analyzed (Participants) | 18 | 18 | 18 | 15 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (6.7) | 65.1 (7.9) | 62.3 (9.3) | 65.1 (7.7) | 64.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 4 | 6 | 31
  Male | 10 | 5 | 14 | 9 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 18 | 18 | 18 | 15 | 69
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Adverse Events Related, Not Related and Serious Events Related to Paracetamol
Description: Phase 1: Number of participants with treatment evaluation and confirmation of the safety of the three doses of paracetamol 3% solution administered in the total number of patients enrolled
Time Frame: In the first 24 hours, in the first 48 hours and at day 7±1
Measure: Number; unit: participants
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL)
Number analyzed (Participants) | 3 | 3 | 3
participants
  Adverse event related | 0 | 0 | 0
  Adverse event not related | 1 | 1 | 6
  Serious adverse event | 0 | 0 | 0

2. Primary Outcome: Phase 2: Pain Intensity
Description: Phase 2: Pain intensity at rest evaluated as VAS scores ( 0-100 mm visual analogue scale : 0 is the absence pain and 100 is the maximum pain sensation)
Time Frame: baseline (0 h), 1, 6, 9, 12, 15, 24, and 48 h after anaesthetic IT injection and at discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 14 | 13 | 15 | 15
units on a scale
  baseline | 11.9 (15.5) | 17.3 (15.6) | 24.5 (19.5) | 10.7 (13.4)
  1 hour after anaesthetic | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  6 hours after anaesthetic | 21.5 (22.2) | 32.2 (25) | 20.3 (25.3) | 42.3 (31.5)
  9 hours after anaesthetic | 21.6 (18) | 13.6 (11.6) | 17.3 (24) | 26.3 (22.3)
  12 hours after anaesthetic | 13.1 (16.5) | 10.1 (8.6) | 11.2 (17.5) | 17.9 (16.7)
  15 hours after anaesthetic | 15.4 (16.7) | 10.2 (10.2) | 10.6 (13.8) | 20.5 (21.5)
  24 hours after anaesthetic | 11.4 (10.7) | 9.5 (8.9) | 13.6 (14.9) | 16 (18.3)
  48 hours after anaesthetic | 6.1 (8.6) | 3.2 (6.6) | 7.7 (12.9) | 8.7 (11.6)
  Discharge | 2.5 (3.7) | 4.1 (4.8) | 4.8 (6.8) | 8.0 (9.6)

3. Secondary Outcome: Phase 2: Morphine
Description: Phase 2: Total morphine use
Time Frame: At 24 and 48 h after anaesthetic IT injection and entire study period, up to 7 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 14 | 13 | 15 | 15
mg
  first 24 hours | 14.1 (10.4) | 12.6 (4.5) | 22.8 (14.7) | 14.3 (7.4)
  first 48 hours | 24.5 (19.7) | 15.8 (5.1) | 33.5 (21.5) | 21 (12.8)
  entire study period | 24.8 (19.7) | 15.8 (5.1) | 33.8 (21.4) | 21.1 (13)

4. Secondary Outcome: Phase 2: Time to First Morphine Use
Description: Phase 2: Time to first morphine use (minutes)
Time Frame: Postoperative, up to 48 hours after end of surgery
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 351 [275 to 503] | 236 [181 to 322] | 318 [184 to 415] | 279 [169 to 313]

5. Secondary Outcome: Phase 2: Number of Participants With Need for Supplemental Analgesia
Description: Phase 2: Need for supplementary analgesia, other than the planned morphine PCA
Time Frame: Postoperative, up to 48 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 9 | 11 | 11 | 10

6. Secondary Outcome: Phase 2: Morphine-related Adverse Events
Description: Percentage of subjects experiencing during the study the morphine-related adverse events pre-specified in the protocol
Time Frame: up to 24 hours after surgery, up to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 1 | 6 | 1 | 6

7. Secondary Outcome: Phase 2: Time to Readiness for Surgery
Description: Time period from completion of spinal injection (time 0 h) to achievement of sensory and motor block adequate for surgery.
Time Frame: Intraoperative
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 9 [5 to 16] | 10 [4 to 10] | 10 [5 to 11] | 8 [5 to 12]

8. Secondary Outcome: Phase 2:Maximum Level of Sensory Block
Description: Sensorial block will be verified by bilateral Pinprick test using a 20-G hypodermic needle and will be recorded. Pinprick sensation will be scored as being present (score 1) or absent (score 0). Onset of sensory block is defined as an absent touch sensation (score 0)
Time Frame: Intraoperative
Measure: Number; unit: participants
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
participants
  T1 | 0 | 0 | 0 | 0
  T2 | 0 | 0 | 0 | 0
  T3 | 0 | 0 | 0 | 0
  T4 | 0 | 2 | 0 | 1
  T5 | 2 | 1 | 0 | 0
  T6 | 4 | 4 | 3 | 3
  T7 | 1 | 2 | 1 | 6
  T8 | 7 | 7 | 10 | 28
  T9 | 0 | 2 | 0 | 2
  T10 | 2 | 0 | 1 | 0
  T11 | 1 | 0 | 0 | 0

9. Secondary Outcome: Phase 2: Time to Sensory Block
Description: Time to maximum level of sensory block
Time Frame: Intraoperative
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 18 [13 to 20] | 15 [9 to 20] | 15 [13 to 20] | 17 [10 to 23]

10. Secondary Outcome: Phase 2: Time to Regression of Spinal Block
Description: Time period from spinal injection (time 0 h) to the time when the Bromage score returns to 0 and sensitive perception returns to S1. Bromage scale:
  I - Free movement of legs and feet II - Just able to flex knees with free movement of feet III - Unable to flex knees, but with free movement of feet IV - Unable to move legs or feet
Time Frame: from readiness for surgery,then every 10 min until the maximum level is reached (two consecutive observations with the same level of sensory block) and then every 30 min until regression of spinal block
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 285 [260 to 345] | 246 [228 to 280] | 265 [245 to 303] | 280 [232 to 302]

11. Secondary Outcome: Phase 2: Vital Signs
Description: Systolic and Diastolic Blood Pressure (mmHg)
Time Frame: at screening, at baseline (before the spinal injection) and at end of the study (Day 6).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
mmHg
  systolic Blood Pressure at screening | 137 (20.4) | 144.6 (20.5) | 148.5 (14.7) | 147.7 (15.7)
  systolic Blood Pressure at baseline | 145.5 (13.6) | 146.3 (19.2) | 138.7 (10.5) | 144.8 (12.3)
  systolic Blood Pressure at end of the study (day6) | 130 (14.6) | 130.3 (11.3) | 133.5 (10.2) | 138.1 (14.5)
  Diastolic Blood Pressure at screening | 87.1 (11.3) | 85.7 (7) | 90.9 (8.2) | 87 (5.1)
  Diastolic Blood Pressure at baseline | 83 (8.8) | 78.9 (10.3) | 77.8 (10) | 85.9 (5.8)
  Diastolic Blood Pressure at end of the study (day6) | 79.5 (10.8) | 78.2 (7.5) | 79 (6.8) | 83.1 (9.3)

12. Secondary Outcome: Phase2: Concomitant Medications
Description: record the concomitant medications intaked during the study
Time Frame: at screening, at baseline until the end of the study (Day 6)
Measure: Number; unit: participants
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
participants
  heparin group | 15 | 15 | 15 | 15
  Second-generation cephalosporins | 15 | 15 | 15 | 15
  Solutions affecting the electrolyte balance | 15 | 15 | 15 | 15
  Direct factor Xa inhibi | 15 | 15 | 14 | 15
  Amino acids | 14 | 13 | 12 | 15
  propofol | 11 | 13 | 13 | 14
  Adrenergic and dopaminergic agents | 10 | 11 | 12 | 12
  Propionic acid derivatives | 7 | 8 | 10 | 6
  Pyrazolones | 4 | 7 | 11 | 9
  Acetic acid derivatives and related substances | 6 | 7 | 8 | 8
  Osmotically acting laxatives | 1 | 3 | 6 | 3
  Proton pump inhibitors | 2 | 4 | 4 | 3
  Serotonin (5HT3) antagonists | 1 | 6 | 2 | 4
  Benzodiazepine derivatives | 2 | 0 | 4 | 2
  ANTIEMETICS AND ANTINAUSEANTS | 1 | 2 | 1 | 3
  Other opioids | 1 | 1 | 1 | 2
  Platelet aggregation inhibitors excl. heparin | 1 | 1 | 0 | 1
  Angiotensin II antagonists, | 1 | 1 | 0 | 0
  Natural opium alkaloids | 0 | 0 | 1 | 1

13. Secondary Outcome: Phase 2: SpO2
Description: Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the blood.
Time Frame: at screening, at baseline (before the spinal injection) and at the end of the study (day 6)
Measure: Mean (Standard Deviation); unit: Oxygen Saturation percentage
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
Oxygen Saturation percentage
  screening | 97.93 (0.59) | 98 (0.53) | 98.27 (0.70) | 97.80 (0.77)
  baseline | 97.27 (1.03) | 97.07 (1.03) | 97.33 (1.18) | 96.87 (1.36)
  end of the study (day 6) | 97.73 (1.03) | 97.53 (0.83) | 97.8 (0.77) | 97.6 (0.74)

14. Secondary Outcome: Phase 2: ECG
Description: Electrocardiography is the process of producing an electrocardiogram (ECG), it is a graph of voltage versus time of the electrical activity of the heart using electrodes placed on the skin.
Time Frame: screening, baseline and end of study (Day 6±1)
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  screening: normal | 10 | 9 | 11 | 11
  screening: Abnormal, Not Clinically Significant | 5 | 6 | 4 | 4
  screening: Abnormal, Clinically Significant | 0 | 0 | 0 | 0
  baseline: normal | 13 | 11 | 11 | 12
  baseline: Abnormal, Not Clinically Significant | 2 | 4 | 4 | 3
  baseline: Abnormal, Clinically Significant | 0 | 0 | 0 | 0
  end of study: normal | 12 | 13 | 11 | 12
  end of study: Abnormal, Not Clinically Significant | 3 | 2 | 4 | 3
  end of study: Abnormal, Clinically Significant | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Clinical study duration (7 days)
Arm/Group | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | 120 mg Paracetamol 3% (4mL) | Phase II Only: Saline Solution 0.9%
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 8/18 | 10/18 | 13/18 | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 mg Paracetamol 3% (2 mL) (N=18) | 90 mg Paracetamol 3% (3 mL) (N=18) | 120 mg Paracetamol 3% (4mL) (N=18) | Phase II Only: Saline Solution 0.9% (N=15)
procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 7 (7) | 3 (3) | 5 (5)
postprocedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 6 (6) | 4 (4)
urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 6 (6) | 3 (3) | 8 (8) | 5 (5)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dyspespsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
epigastric disconfrort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
prupritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
antiementic supportive care (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT02654860/Prot_SAP_000.pdf